CLINICAL TRIAL: NCT02207803
Title: A Culturally Sensitive Intervention for TBI Caregivers in Latin America
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HM20001660; R21TW009746 (NIH)
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-09

CONDITIONS: Traumatic Brain Injury
Keywords: Brain Injuries; Caregivers; Intervention Studies; Latin America
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Experimental Transition Assistance Program
  Interventions: Behavioral: Transition Assistance Program
- Control (No Intervention): Control

INTERVENTIONS:
Behavioral: Transition Assistance Program
  Arms: Intervention

SUMMARY:
Traumatic brain injury (TBI) patients in Latin America experience high levels of disability and extremely poor functional outcomes, and their informal caregivers play a key role in their rehabilitation and care. To improve TBI rehabilitation through stronger informal caregiving, the proposed study will develop and evaluate an evidence--based and culturally sensitive Transition Assistance Program for informal caregivers of patients with TBI in Latin America during the patient's transition from hospital to home. This study will generate findings that can provide empirically supported guidance to clinicians regarding the provision of culturally tailored rehabilitation services for TBI caregivers in Latin America and in the U.S.

ELIGIBILITY:
TBI Patient Inclusion Criteria:

* Will be discharged home and not to a nursing home
* Give permission for their caregiver to participate
* Sign an informed consent
* Have the ability to communicate over the phone for data collection
* Are between 18-60 years of age

Caregiver Inclusion Criteria

* Have a telephone in the home or cellular phone and are able to talk on the phone
* Sign an informed consent
* Score at least a 13 on a health literacy screening tool
* Are between 18-85 years of age

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-01; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul B. Perrin, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (3):
- Colombia (2):
  - Pontificia Universidad Javeriana Cali, Cali
  - Universidad Sur Colombiana, Neiva
- National Institute of Neurology and Neurosurgery, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Transition Assistance Program: Group receiving the 5-session behavioral treatment from a clinician
- Control: Group receiving the standard of care at the rehabilitation facility
Period: Overall Study
Arm/Group | Transition Assistance Program | Control
Started | 125 | 125
Completed | 110 | 108
Not Completed | 15 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transition Assistance Program | Control | Total
Number analyzed (Participants) | 125 | 125 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 120 | 119 | 239
  >=65 years | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37 (14) | 39 (13) | 38 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 63 | 124
  Male | 64 | 62 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 125 | 125 | 250
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Colombia | 44 | 44 | 88
  Mexico | 81 | 81 | 162

OUTCOME MEASURES:

1. Primary Outcome: Zarit Burden Interview
Description: 22-item measure of caregiver self-reported burden. Response options for each item range from 0-4, and total scores range from 0-88, with higher scores indicating greater self-reported burden. Only total scores are reported here.
Time Frame: 2 months post-hospital discharge
Population: Data are from caregivers only, hence not the full sample.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transition Assistance Program | Control
Number analyzed (Participants) | 56 | 56
units on a scale | 23.41 (16.50) | 26.48 (19.71)

2. Secondary Outcome: Exemplary Care Scale-Provide Subscale
Description: 4-item measure of the patient's report of the quality of care they receive from their caregiver. Response options for each item range from 1-4, and total scores range from 4-16, with higher scores indicating a higher quality of informal care received. Only Provide subscale scores of the Exemplary Care Scale are reported here.
Time Frame: 2 months post-hospital discharge
Population: This is patient-report only at post-test, hence it does not use the full sample.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transition Assistance Program | Control
Number analyzed (Participants) | 56 | 56
units on a scale | 14.23 (2.89) | 14.07 (2.64)

ADVERSE EVENTS:
Time Frame: 4-month data collection window
Arm/Group | Transition Assistance Program | Control
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/125
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/125
Other Adverse Events (participants affected / at risk) | 0/125 | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-05-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT02207803/SAP_000.pdf
  • Study Protocol (2014-05-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT02207803/Prot_001.pdf